CLINICAL TRIAL: NCT00805376
Title: Phase I Trial of Conditionally Replication-Competent Adenovirus (DNX-2401, Formerly Known as Delta-24-RGD-4C) for Recurrent Malignant Gliomas
Brief Title: DNX-2401 (Formerly Known as Delta-24-RGD-4C) for Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DNAtrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-310
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-01

CONDITIONS: Brain Cancer; Central Nervous System Diseases
Keywords: Brain; Brain Cancer; Central Nervous System Diseases; CNS; Conditionally Replication-Competent Adenovirus; Delta-24-RGD; DNX-2401; Recurrent Malignant Gliomas; malignant brain tumor
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Diseases; Glioma | interventions — Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: DNX-2401 (Experimental): Surgical procedure precisely injects DNX-2401 through a catheter (small tube) into brain tumor.
  Interventions: Drug: DNX-2401
- Group B: DNX-2401 + Surgery (Experimental): DNX-2401 injection + Tumor removal
  Interventions: Drug: DNX-2401; Procedure: Tumor Removal

INTERVENTIONS:
Drug: DNX-2401 — Surgical procedure precisely injects DNX-2401 through a catheter (small tube) into brain tumor.
  Other Names: Delta-24-RGD-4C
Procedure: Tumor Removal — Surgical Tumor Resection
  Other Names: Craniotomy
  Arms: Group B: DNX-2401 + Surgery

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of DNX-2401 that can be injected directly into brain tumors and into the surrounding brain tissue where tumor cells can multiply. A second goal is to study how the new drug DNX-2401 affects brain tumor cells and the body in general.

DETAILED DESCRIPTION:
The Study Drug:

DNX-2401 (formerly known as Delta-24-RGD-4C) is a virus that works by killing brain tumor cells. It is made from a common cold virus, called adenovirus, type 5. This virus normally causes the common cold, and most people around the world have been exposed many times to this common, naturally-occurring virus during their lives. Two (2) changes have been made to the adenovirus to make DNX-2401. The first change was to make the virus only grow in cancer cells. The second change was made to allow DNX-2401 to enter cancer cells more easily. These changes make DNX-2401 more able to multiply and kill cancer cells and less likely to multiply in normal cells.

Study Groups:

Participants will eventually be divided into 2 groups (Groups A and B).

At first, all participants will only be enrolled into Group A. Participants in Group A will receive the study drug but will not have the recurrent malignant glioma tumor removed by surgery.

Enrollment into Group B will not start until the FDA has reviewed initial results on how the treatment for participants in Group A effected brain tumor cells and the body in general. Once approval for enrollment is given, all eligible participants will be assigned to Group B and will receive the study drug and have their tumors removed by surgery. If you are to receive surgery, you will be asked to sign a separate surgical consent form to help further explain the operation.

If you are found to be eligible to take part in this study, you will be assigned to a dose level of DNX-2401 based on when you joined this study. Up 8 dose levels of DNX-2401 will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of DNX-2401 is found. You will be informed of which dose you will receive.

Study Drug Administration:

DNX-2401 is given by a surgical procedure where a neurosurgeon precisely injects DNX-2401 through a catheter (small tube) that is inserted into your brain tumor. You will stay in the hospital and be watched closely afterward for up to 48 hours, but it may be longer if your doctors feel that you are not ready to go home.

After receiving DNX-2401, all participants must wear a mask. You must also stay away from pregnant women, babies, children under three years of age, elderly people and large groups of people who may have weaker defenses to disease or those who can spread a disease. You must also stay away from other patients who may have immune system problems, such as people with AIDS, or people who are getting chemotherapy or radiation therapy. The study doctors will decide how long you will need to follow these precautions. You should not donate blood or sperm for at least 6 months after receiving DNX-2401.

Group A:

Before receiving DNX-2401, participants in Group A will have a sample (stereotactic biopsy) of brain tumor tissue collected to confirm that recurrent malignant glioma is present. On the morning of the biopsy, you will have an MRI (with dye). A metal frame will be placed on your head and an MRI of your brain will be done. Before the MRI, a dye will be injected to help give the doctors a better picture of your brain. The head frame allows the surgeon to use MRI to identify the precise location of the tumor within the brain. The frame will stay in place for several hours while the procedure is being performed.

A portion of your head will be shaved for the biopsy. You will have a small incision (cut) in your head (about 2-3 inches). The protective covering of the brain (dura) will be opened and a piece of brain tumor will be removed. If, under a microscope, the biopsy shows that the tumor is still malignant glioma, you will then have an injection of DNX-2401. The anesthesiologists (doctor who gives the anesthesia) may give you medication to make you sedated (anesthesia). They will place a needle into your vein (intravenous line or "IV") to give you this medicine. The anesthesia is given so that you do not feel any pain or discomfort and do not move during the MRI or the surgery.

A small catheter will be placed into the tumor and the metal frame will help guide the proper placement. Some anti-inflammatory medication (a steroid called dexamethasone) will be given in your vein. Then DNX-2401 will be slowly injected into the tumor over about 10 minutes. After the injection, the incision will be closed in a standard and cosmetically acceptable manner.

Group B:

Before receiving DNX-2401, participants in Group B will have a biopsy to confirm that the tumor is recurrent glioma. The procedure will be exactly the same as described for those in Group A. This is called "Stage 1." However, at the end of the biopsy and study drug injection procedure, the catheter will be clipped off next to your skull and a portion of the tube will remain inside the tumor and in place for the next 2 weeks. The scalp will be closed over the clipped catheter to prevent any possibility of infection. The next day, you will have a CT scan to check the tumor and placement of the catheter.

Group A Follow-up Visits:

You will come back to the study center for check-ups at 4, 7,14 and 28 days, then 2, 3, and 4 months after the injections, and then every 2 months for 2 years. After that, you will be asked to return to the clinic every 4 months for the rest of your life. At each visit, the following tests and procedures will be performed:

* You will be asked to give information about any new medications and therapies, including vitamins, herbs, and supplements that you may be taking.
* You will be asked to describe any changes in your health or how you feel.
* You will have a neurological exam.
* Your weight will be measured on Day 28 and at 2, 3 and 4 months.
* Your vital signs will be measured.
* You will be asked to provide a blood sample (about 1 teaspoon), a urine sample and a swab of your nose and throat will be taken.
* You will have blood tests (about 4 teaspoons) to evaluate your clinical status on Days 4, 7, 28, and at 2, 3 and 4 months.
* Blood (about 2 teaspoons) will be collected to look for the presence of anti-AD5 and virus.
* Women who are able to become pregnant must have a blood (about 1 teaspoon) pregnancy test on 1 and 4 month visit and all follow-up visits after that.
* You will have an MRI at each visit except for Day 4.
* After the 4 month visit, you will have an evaluation to see how you have responded to treatment for the first 2 years and every 4 months after that.

Group B Follow-up Visits:

You will be seen in the study center for check-ups on Days 4, 7, and 13 after the injection but before your craniotomy. At each visit the following tests and procedures will be performed:

* You will be asked to give information about any new medications and therapies, including vitamins, herbs, and supplements that you may be taking.
* You will be asked to describe any changes in your health or how you feel.
* You will have a neurological exam.
* Your vital signs will be measured.
* You will be asked to provide a blood sample (about 1 teaspoon), a urine sample and a swab of your nose and throat will be taken.
* You will have a blood test (about 4 teaspoons) to evaluate your clinical status.
* Blood (about 2 teaspoons) will be collected to look for the presence of anti-AD5 and virus.
* Women who are able to become pregnant must have a blood (about 1 teaspoon) pregnancy test on Day 13, 1 and 4 month visits and all follow-up visits after that.
* You will have an MRI on Days 7 and 13 only.

If you are feeling well 14 days after the first injection of study drug, you will be brought back to the operating room for a second procedure to remove the tumor. You will undergo a craniotomy, in which the skull over the tumor is removed to get to the brain and tumor. The neurosurgeon will try to remove the tumor as completely as possible with the catheter tip from the first procedure in place. After the tumor has been removed, you will receive another dose of DNX-2401 that will be injected into the brain tissue that surrounded the tumor to try to kill any remaining tumor cells. This is called "Stage 2." The skull will then be replaced and the skin closed. Within 6 hours of the craniotomy on Day 14, you will have a neurological exam and your vital signs will be measured.

On the day of resection, a sample of the removed brain tumor tissue will be collected and stored until the study is over. Analysis of the tissue will be performed to look for the presence and activity of the virus, as well as any additional tests that are necessary for protocol purposes.

Group B Follow-up Visits after Craniotomy:

After the surgery, you will be seen in the hospital or come back to the center on Days 15, 18, 21, 28, and 42, at 2, 3 and 4 months, and then every 2 months for 2 years. After that, you will be asked to come back every 4 months for the rest of your life. At each visit, the following tests and procedures will be performed:

* You will be asked to give information about any new medications and therapies, including vitamins, herbs, and supplements that you may be taking.
* You will be asked to describe any changes in your health or how you feel.
* You will have a neurological exam.
* Your weight will be measured on Day 28, 42 and at 2, 3 and 4 months only.
* Your vital signs will be measured.
* You will be asked to provide a blood sample (about 1 teaspoon), a urine sample, and a swab of your nose and throat.
* You will have a blood test (about 4 teaspoons) to evaluate your clinical status.
* Blood (about 2 teaspoons) will be drawn to look for the presence of anti-AD5 and virus.
* Women who can become pregnant must have a blood (about 1 teaspoon) pregnancy test at all visits except Day 15 and 18.
* You will have an MRI.

For participants who are clinically unable to wait 14 days for surgery because of the tumor's size and/or location, or because they are experiencing serious neurological symptoms, the study chair may decide to skip the biopsy.

Group B Follow-up Visits (Stage 2--Craniotomy Only):

After the surgery, you will be seen in the hospital or come back to the center on Days 1, 4, 7, 14, and 28; at 2, 3, and 4 months; and then every 2 months for 2 years. After that, you will be asked to come back every 4 months for the rest of your life. At each visit, the following tests and procedures will be performed:

* You will be asked to give information about any new medications and therapies, including vitamins, herbs, and supplements that you may be taking.
* You will be asked to describe any changes in your health or how you feel.
* You will have a neurological exam.
* Your weight will be measured on Day 28 and at 2, 3, and 4 months.
* Your vital signs will be measured.
* You will be asked to provide a blood sample (about 1 teaspoon), a urine sample, and a swab of your nose and throat.
* You will have a blood test (about 4 teaspoons) to evaluate your clinical status.
* Blood (about 2 teaspoons) will be drawn to look for the presence of anti-AD5 and virus.
* Women who can become pregnant must have a blood (about 1 teaspoon) pregnancy test on 1- and 4-month visit and all follow-up visits after that.
* You will have an MRI.

This is an investigational study. At this time, DNX-2401 is only being used in research. Up to 96 patients will take part in this study (up to 48 in Group A and 48 in Group B). All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven recurrent malignant primary glioma will be eligible. Glioma type will be restricted to: GBM, gliosarcoma (GS), anaplastic gliomas [anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic infiltrating glioma (AIG), mixed anaplastic glioma (MAG), anaplastic ependymoma]
2. Patients must show unequivocal evidence for tumor recurrence or progression by MRI scan within 15 days prior to Day 0/Baseline procedure after failing prior surgical resection, biopsy, chemotherapy or radiation
3. For patients entered in Group A (see Treatment Plan) tumors must be accessible for stereotactic injection. Tumors must be between 1.0 - 5.0 cm in diameter
4. For patients entered in Group B (see Treatment Plan) tumors must be surgically resectable, and surgical resection must be indicated at the time of baseline evaluation. Tumors must be >1.0 cm in diameter.
5. Patients will consent to have a biopsy taken at the time of the stereotactic injection to confirm the presence of malignant glioma (based on frozen section) before injection of DNX-2401
6. For each patient there must be a consensus between the physician investigators in this study that injection will not deliver DNX-2401 into the ventricular system. Patients must have a stable steroid regimen for at least 1 week prior to DNX-2401 administration
7. Patients may or may not have had prior chemotherapy
8. Patients must be willing and able to give informed consent
9. Age > /= 18 years
10. Patients must have a Karnofsky performance status greater than or equal to 70
11. Patients must have recovered from the toxic effects of prior therapy (i.e., CTC grade 1 or less). For example, they must be at least two weeks after vincristine, 6 weeks after nitrosoureas, and 3 weeks after procarbazine or temozolomide administration
12. Patients must have adequate bone marrow function (absolute granulocyte count > 1,500 and platelet count of > 100,000), adequate liver function (SGPT and alkaline phosphatase < 2 times institutional normals and bilirubin <1.5 mg%), and adequate renal function (BUN or creatinine <1.5 times institutional normal) prior to starting therapy
13. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender
14. No exclusion to this study will be based on race. Minorities will actively be recruited to participate. The malignant glioma patient population treated at MDACC over the past year is as follows: American Indian or Alaskan Native - 0, Asian or Pacific Islander - <2%, Black, not of Hispanic Origin - 3%, Hispanic - 6%, White, not of Hispanic Origin - 88%, Other or Unknown - 2%, Total - 100%

Exclusion Criteria:

1. Any radiotherapy within 4 weeks prior to date of DNX-2401 administration.
2. Active uncontrolled infection or severe intercurrent medical conditions. All patients must be afebrile at baseline (i.e., < 38.0 Celsius [C])
3. Evidence of bleeding diathesis or use of anticoagulant medication or any medication that may increase the risk of bleeding that cannot be stopped prior to surgery. If the medication can be discontinued , based on the clinical judgment of the surgeon, prior to DNX-2401 injection then patient may be eligible.
4. History or current diagnosis of any medical or psychological condition that in the Investigator's opinion, might interfere with the subject's ability to participate or inability to obtain informed consent because of psychiatric or complicating medical problems
5. Female who is pregnant and/or nursing. Because of the potential risk of a recombinant virus containing a gene involved in cellular growth regulation and differentiation which could potentially affect a developing fetus or growing infant, females who are pregnant, at risk of pregnancy, or breast feeding a baby during the study period are excluded
6. Tumor position that, in the Investigator's opinion, would pose the risk of penetration of the cerebral ventricular system during injection with study drug. If, during the DNX-2401injection procedure, penetration of the ventricular system is suspected or confirmed, DNX-2401 administration will be aborted
7. Immunocompromised subjects, subjects with autoimmune conditions, active hepatitis (B or C) or HIV seropositivity
8. Patients with Li-Fraumeni Syndrome or with a known germ line deficit in the retinoblastoma gene or its related pathways
9. Multiple intracranial malignant glioma lesions at the time of recurrence. Multiple enhancing areas within a single tumor will not be considered multiple glioma lesions
10. Tumor involvement which would require ventricular, brainstem or posterior fossa injection or access through a ventricle in order to deliver the virus
11. Tumor involving the subependyma or suspected cerebrospinal fluid (CSF) dissemination
12. Documented extracranial metastasis
13. Biologic/immunotherapy (e.g., IL-2, IL-12, interferon) within 4 weeks of DNX-2401 administration
14. Concurrent chemotherapy, radiation or biological therapy
15. Any contraindication for undergoing MRI such as: individuals with pacemakers, epicardial pacer wires, infusion pumps, surgical and/or aneurysm clips, shrapnel, metal prosthesis, implants with potential magnetic properties, metallic bodies in the eyes, etc.
16. White blood cell (WBC) < 2.5 x 103/mm3, absolute neutrophil count (ANC) < 1.5 x 103/mm3, platelet < 100,000/mm3, hemoglobin (Hgb) < 10.0 gm/dL, prothrombin time/international normalized ratio (PT/INR) or partial thromboplastin time (PTT) > 1.8 x control
17. Grade 4 hematological toxicity
18. Serum creatinine > 1.5 mg/dL
19. Liver transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) or total bilirubin > 2x the upper limits of normal
20. Vaccinations of any kind within 30 days prior to Delta-24-RGD-4C administration
21. Current diagnosis of other cancer except curative cervical cancer in situ, basal or squamous cell carcinoma of the skin. Patients with a history of another cancer, but who are cancer free for a minimum of three years remain eligible
22. History of encephalitis, multiple sclerosis, other CNS infection or primary CNS disease that would interfere with subject evaluation
23. Patients with history of prior gene transfer therapy or prior therapy with cytolytic virus of any type, especially DNX-2401
24. Males or females who refuse to use a double-barrier form of birth control during the study and for up to 6 months after injection with DNX-2401

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) DNX-2401 | Assessed during 14 day waiting period between doses (every 28 days).
  Each cohort of three subjects each sequentially assigned to escalating doses of DNX-2401, with acceptable grade of neurotoxicity Common Toxicity Criteria (CTC) < grade 3, related to the study drug, and according to standard Gehan phase I dose-escalating criteria for toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick F. Lang, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lang FF, Conrad C, Gomez-Manzano C, Yung WKA, Sawaya R, Weinberg JS, Prabhu SS, Rao G, Fuller GN, Aldape KD, Gumin J, Vence LM, Wistuba I, Rodriguez-Canales J, Villalobos PA, Dirven CMF, Tejada S, Valle RD, Alonso MM, Ewald B, Peterkin JJ, Tufaro F, Fueyo J. Phase I Study of DNX-2401 (Delta-24-RGD) Oncolytic Adenovirus: Replication and Immunotherapeutic Effects in Recurrent Malignant Glioma. J Clin Oncol. 2018 May 10;36(14):1419-1427. doi: 10.1200/JCO.2017.75.8219. Epub 2018 Feb 12. PMID 29432077